CLINICAL TRIAL: NCT05326386
Title: Gamification and Social Incentives to Augment Medication Adherence
Brief Title: Gamification and Medication Adherence (GAME Adherence)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 850287
Record Dates: First submitted 2022-03-21; First posted 2022-04-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypertension and Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Via the Way to Health platform, all participants will receive daily text messages asking about medication adherence for that day and twice weekly text messages asking if participants have measured blood pressure on that day.
- Intervention (Experimental): Via the Way to Health platform, all patients will receive daily text messages asking about medication adherence for that day and twice weekly text messages asking if participants have measured blood pressure on that day.
  Participants are entered into a game. Each week they receive 90 points. If they took their medications or checked their blood pressure the prior day, they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 70 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner. At the start of the intervention, the study team holds a 3-way phone call with the participant and support partner to discuss ways they can help the participant meet their goal. The support partner gets a weekly email with the participant's progress.
  Primary care physicians will receive a monthly email noting patients' self-reported adherence and blood pressure.
  Interventions: Behavioral: HTN and Medication Adherence

INTERVENTIONS:
Behavioral: HTN and Medication Adherence — Via the Way to Health platform, all patients will receive daily text messages asking about medication adherence for that day and twice weekly text messages asking if participants have measured blood pressure on that day.
  Participants are entered into a game. Each week they receive 90 points. If they took their medications or checked their blood pressure the prior day, they keep their points, but if not, they lose 10 points. At the end of the week if they have at least 70 points they move up a level, but if not, they drop a level. Participants start in the middle of 5 levels.
  Participants choose a support partner. At the start of the intervention, the study team holds a 3-way phone call with the participant and support partner to discuss ways they can help the participant meet their goal. The support partner gets a weekly email with the participant's progress.
  Primary care physicians will receive a monthly email noting patients' self-reported adherence and blood pressure.
  Arms: Intervention

SUMMARY:
A two-arm randomized controlled trial to evaluate whether a gamification intervention plus involvement of a supportive partner (social support) and sending reports to physicians (accountability) increases medication adherence in patients with hypertension and hyperlipidemia. The study will randomize 84 patients with hypertension, hyperlipidemia, and a history of poor medication adherence seen in a single Penn Medicine clinic to an 18-week gamification intervention or to attention control text messages alone.

DETAILED DESCRIPTION:
Atherosclerotic cardiovascular disease (ASCVD) is the leading cause of morbidity and mortality in the United States. Hypertension and hyperlipidemia have been recognized as risk factors for ASCVD for more than 60 years, with several low-cost medications approved for treatment offering up to 88% reduction of cardiovascular events with perfect adherence. Poor medication adherence is an important contributor to poor risk factor control, and affects Black patients and those with low socioeconomic status to a greater extent than other populations. Interventions specifically targeting improved medication adherence in Black communities and those with low socioeconomic status may therefore improve cardiovascular health in these vulnerable groups. Previous trials have used multiple different methods to increase medical adherence, but few of these methods have been implemented due to their high cost and/or personnel-heavy approaches. Leveraging insights from behavioral economics may facilitate a lower touch, less expensive, and ultimately more scalable approach to increase medication adherence. Therefore, the investigators will perform a randomized controlled trial of a gamification intervention that leverages insights from behavioral economics-based versus attention control to determine the effect of the gamification intervention on medication adherence. Participants will include patients with poorly-controlled hypertension, hyperlipidemia, and a history of nonadherence to medications from a single clinic that serves patients from West and Southwest Philadelphia, a community with a high proportion of Black individuals. Patients in both arms will be provided with a blood pressure cuff and enrolled in an automated bidirectional text messaging platform that will send daily texts asking about medication adherence and twice weekly texts asking if participants have measured their blood pressure that day. The intervention arm will include a precommitment pledge, weekly progression (or regression) through levels with loss-framing of points, support from a family member or friend, and accountability from a primary care physician. After 18 weeks, changes in patient-reported medication adherence (primary outcome) will be compared between study arms along with patient-reported blood pressure and medication possession ratio (MPR).

ELIGIBILITY:
Inclusion Criteria:

* Prescribed 1 or 2 blood pressure medications and a statin medication for > 1 year
* Has supply of medications at the time of enrollment
* Medication possession ratio 40-80% for at least one of those medications for the past 6 months
* Systolic blood pressure > 140 mm Hg at most recent check
* Owns a smartphone or tablet operating the iOS or Android operating system

Exclusion Criteria:

* Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension of English)
* Systolic blood pressure > 180 mm Hg at their last bp check
* Anticipated life expectancy less than 6 months
* Any other reason why it is not feasible to complete the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
patient-reported adherence | 18 weeks
  Patient reported adherence will be defined as days taking all prescribed antihypertensive medications and statins divided by total days in the study over the entire study duration; this will be compared between study arms

SECONDARY OUTCOMES:
Change in blood pressure over study duration | 18 weeks
  Patients will measure their systolic and diastolic blood pressure twice weekly using a blood pressure cuff provided by the study and report the values via text message. We will compare change in systolic and diastolic blood pressure from study start to the end of the study between intervention and control arms
Patient-reported adherence in weeks 14-18 | 5 weeks (during study weeks 14-18)
  Patient reported adherence will be defined as days taking all prescribed antihypertensive medications and statins divided by total days in the study during study weeks 14-18; this will be compared between study arms.
Medication possession ratio over study duration | 18 weeks
  Medication possession ratio will be calculated as the number of days that a patient has a supply of medication divided by the total number of days in the study; this will be compared between arms
Medication possession ratio in weeks 14-18 | 5 weeks (during study weeks 14-18)
  Medication possession ratio will be calculated as the number of days that a patient has a supply of medication divided by the total number of days in the study from weeks 14-18; this will be compared between arms

OTHER OUTCOMES:
Change in low density lipoprotein cholesterol | 18 weeks
  At the end of the study, participants will have their low density lipoprotein cholesterol checked. We will compare the change from baseline to follow-up LDL between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States